CLINICAL TRIAL: NCT00548522
Title: Pancreatic Islet Mass in Pregnancy - Pilot Study
Brief Title: Pancreatic Islet Mass in Pregnancy in Type 1 Diabetes
Status: Terminated | Type: Observational
Why Stopped: Difficulty in finding staff to help with study
Sponsor: University of Alberta (Other)
Responsible Party: Principal Investigator, Edmond A Ryan, Professor, University of Alberta
Other Study IDs: UAHREB4503
Record Dates: First submitted 2007-10-23; First posted 2007-10-24 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-05

CONDITIONS: Type 1 Diabetes; Pregnancy
Keywords: Type 1 Diabetes; Pregnancy; Islet Mass; C-peptide
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Plasma Samples kept for batching of antibody assays
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- 1: Pregnant (12 - 16 wks gestation) women with Type 1 diabetes
- 2: Pregnant women (34-38 wks gestation) with Type 1 diabetes
- 3: Post partum women with Type 1 diabetes
- 4: Non pregnant women with Type 1 diabetes

SUMMARY:
Type 1 diabetic women have a decrease in insulin requirements during early pregnancy. Preliminary evidence suggests this decrease may be secondary to the regeneration of pancreatic B-cells during pregnancy During the second and third trimesters, insulin requirements in Type 1 diabetic women progressively increase until approximately 36 weeks gestation at which time there is a plateau, and frequently, a drop in insulin requirements. We hypothesize that there is regeneration of pancreatic islet cell mass in Type 1 diabetic women during pregnancy. In a cross-sectional study, we will use the acute insulin c-peptide response to arginine to determine if pancreatic islet mass increases at 12 and 36 weeks gestation. Type 1 diabetic women who are not pregnant, who are at 12 and 36 weeks gestation, and who are 6 weeks post-partum will undergo an intravenous arginine tolerance test following an overnight fast. If we find that there is regeneration of beta cells it opens the possibility that therapy may be directed to the same end for people with Type 1 diabetes.

DETAILED DESCRIPTION:
For the pilot phase of this study we will contact women with type 1 diabetes. The study will be explained and the subjects will be asked to sign an informed consent. Each subject will be asked to complete a brief medical history and lifestyle questionnaire.

Subjects will have blood samples taken for glucose and C-peptide and an intravenous arginine stimulation test. For the study tests, subjects will be asked to come to the Clinical Investigations Unit at the University of Alberta Hospital after an overnight fast only once during the study. The intravenous arginine test is a 10 minute test and does not cause hyperglycemia, an advantage over glucose in the setting of pregnancy.

Arginine infusion The intravenous arginine infusion test will be performed after an overnight fast greater than or equal to 8 hours. Subjects may drink water. For the Type 1 diabetic patients on insulin, long-acting insulin may be taken no less than 8 hours prior to the test; no food or short-acting insulin may be taken within 5 hours of the test. Lispro insulin should not be taken within 4 hours of the test.

On the morning of the test, an intravenous catheter, using a 20 gauge IV intercath, will be placed in an antecubital vein in one arm both for sampling and for infusion. Veins will be kept patent with an infusion of NaCl (0.9%) at 25 mL/hr throughout the test. The arm from which samples are obtained will be warmed to 55 C with a heating blanket to assist in the arterialization of the venous samples.

Baseline blood samples for glucose and C-peptide measurements will be drawn in a serum gel barrier tube at minus 10 and 0 minutes. An injection of 5 g of arginine (20 ml Sabex) diluted with 20 ml normal saline to equal 40 ml will be administered over 30 seconds, starting at time 0. The vein will immediately be flushed with 20mL normal saline. Blood samples for insulin and C-peptide will be drawn in barrier tubes at 2, 3, 4, 5, 7 and 10 minutes and serum will be separated and transferred into a cryogenic tube for analysis.

The acute C-peptide response to arginine is defined as the mean of the three highest insulin or C-peptide values between 2 and 5 minutes after the start of the arginine infusion with the mean of the minus 10 and 0 values subtracted.

Blood samples (basal and stimulated) will be analyzed for glucose and C-peptide. The insulin response will not be measured in these Type 1 subjects as it would be meaningless and the C-peptide response will be used.

Blood glucose will be determined by the hexokinase method using the Hitachi 917 system (Roche Diagnostics, Indianapolis, IN).

C-peptide assay An Ultrasensitive C-peptide ELISA method will be used to analyze for C-peptide. This test is specific for low concentrations of C-peptide in blood, specifically for patients with abnormal insulin secretion.

Statistical Analysis/Power calculation

Upon the significance test results for group differences, we will proceed with multiple comparisons of groups to locate the source of significance, while adjusting for multiple significance testing, using the method of Bonferroni.

Expected Possible Findings/ Conclusion

We hope to show that pancreatic islet mass may be present in women with Type 1 diabetes. Any demonstration of beta-cell recovery even in the unique setting of pregnancy would be exciting, as it would demonstrate progenitor beta cells present in the pancreas in type 1 diabetes subjects.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* Females with Type 1 diabetes for at least 5 years
* Diabetes onset < 21 years
* Lean at diabetes onset
* Insulin required from diagnosis
* Willing to undergo intravenous arginine tolerance tests

Exclusion Criteria:

* Inability to provide informed consent
* Any medical condition that would preclude safe conduct of the intravenous arginine
* A family history which includes three generations of family members with the diagnosis of diabetes mellitus
* Women with elevated serum creatinine as arginine is excreted by the kidneys.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Pregnant women with Type 1 diabetes
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2007-08; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
The documentation of Cpeptide in women with type 1 diabetes who are pregnant | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Edmond A Ryan, MD, Principal Investigator — University of Alberta
Locations (2):
- Canada (2):
  - University of Alberta Hospital, Edmonton, Alberta
  - University of Alberta, Edmonton, Alberta